CLINICAL TRIAL: NCT01939262
Title: The Impact of Dietary Restriction of Animal Protein and Fat on Subjective Complaints of Osteoarthritis
Brief Title: The Impact of Dietary Restriction of Animal Protein and Fat on Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essentia Health (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Mary Clifton, Medical Doctor, Essentia Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Osteoarthritis Diet
Record Dates: First submitted 2013-09-05; First posted 2013-09-11 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Osteoarthritis
Keywords: Arthritis; Pain; Function; Diet; Vegan; Vegetarian; Restriction
MeSH Terms: conditions — Osteoarthritis; Arthritis; Pain | interventions — Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vegan Diet (Experimental): Limitation of Animal Fat and Protein in the Diet. Animal products were proscribed and the use of unrefined foods was encouraged. Participants were asked to limit high-fat plant foods, such as nuts, avocados, and refined oils. There was no restriction in energy intake, were encouraged to eat freely and not count calories.
  Interventions: Other: Limitation of Animal Fat and Protein in the Diet
- Control (Placebo Comparator): Subjects maintained their existing diet without modification.
  Interventions: Other: Control

INTERVENTIONS:
Other: Limitation of Animal Fat and Protein in the Diet — Animal products were proscribed and the use of unrefined foods was encouraged. Participants were asked to limit high-fat plant foods, such as nuts, avocados, and refined oils. There was no restriction in energy intake, were encouraged to eat freely and not count calories.
  Arms: Vegan Diet
Other: Control — Participants assigned to the control group will be instructed to follow their usual diets.
  Arms: Control

SUMMARY:
Patients will be randomized into the control or intervention group. Based on patient preference, the intervention group will be trained for one hour in either individual or group format on vegan diet. They will also be directed to www.pcrm.org and www.drmarymd.com for low glycemic, animal free, low fat food options and support. The control group will continue their normal omnivorous diet program. Twenty-four hour food recalls will be obtained at the start and end of the trial, and once a week for the 6 weeks of the trial by telephone. Patients will undergo a final interview at the end of the 6 week study period. The intervention group should strive to obtain 90% of their calories from plants. They will be encouraged to eat freely and not count calories. Patients will undergo additional individual consultation as needed to promote compliance and answer specific questions.

Over the 6 weeks, the Patient Global Improvement of Change (PGIC) and the 36 item short form health survey (SF-36) will be performed weekly by telephone. Patient will perform a Visual Analog Scale (VAS) of their pain level randomly daily on their own. C-reactive protein levels will be assessed at the beginning and end of the study at Munson Medical Center Laboratories as a secondary measure of diet changes.

There have been no published prospective randomized controlled trials assessing whether a vegan diet would benefit osteoarthritis. The specific aim of this study is to determine if a vegan diet will result in subjective reduction in perceived pain and limitations to function in patients with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling
* Medical Provider diagnosis of Osteoarthritis

Exclusion Criteria:

* Pre-existing vegans or vegetarians
* Ages less than 18 or greater than 70
* History of an eating disorder
* History of diabetes
* Inability to afford food
* Lack of control over the food eaten
* Pregnant or nursing
* Known food allergies
* Patients following a medically prescribed diet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Subjective Complaints of Pain and Functionality in Osteoarthritis Patients | Six weeks
  Significant responders were defined as patients that experienced a clinically significant improvement in at least two of the three administered tests: pain, as measured by a 30% improvement on the VAS(Visual Analog Scale) and improvement in patient's global status, measured by a rating of somewhat better to a great deal better on the PGIC scale, and physical function, a >6 point improvement on the 36-item short form health survey (SF-36v2) Role Physical or Physical Component Summary Score

SECONDARY OUTCOMES:
c-reactive protein | 6 weeks
  Clinical laboratory tests of c-reactive protein was drawn at the intake and exit of the study .

CONTACTS AND LOCATIONS:
Overall Officials: Mary R Clifton, MD, Principal Investigator — Essentia Health
Locations (1):
- Mary R Clifton, MD (private solo practice office), Traverse City, Michigan, United States